CLINICAL TRIAL: NCT06660069
Title: A 12-Week, Randomised, Controlled, Examiner-blind, Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste With a Cetylpyridinium Chloride Mouthwash in Improving Gingival Health and Reducing Plaque Accumulation
Brief Title: A Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste With a Cetylpyridinium Chloride Mouthwash in Improving Gingival Health and Reducing Plaque Accumulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 300211
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toothpaste/Mouthwash (SnF2 Toothpaste followed by CPC Mouthwash) (Experimental): Participants will brush their teeth with full ribbon of test toothpaste containing SnF2 on head of toothbrush provided for at least one (timed) minute twice daily (morning and evening) for 12 weeks. After each brushing, participants will swish 20 milliliters (mL) of the mouthwash containing CPC vigorously between teeth for 30 seconds twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Stannous Fluoride Toothpaste (Parodontax Complete Protection Toothpaste); Drug: CPC Mouthwash (Parodontax Active Gum Health Mouthwash)
- Negative Control Toothpaste (Sodium Fluoride Toothpaste) (Active Comparator): Participants will brush their teeth with full ribbon of negative control toothpaste containing sodium fluoride on head of toothbrush provided for at least one (timed) minute twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Regular Fluoride Toothpaste (Crest Cavity Protection)
- Reference Toothpaste (SnF2 Toothpaste) (Active Comparator): Participants will brush their teeth with full ribbon of reference toothpaste containing SnF2 on head of toothbrush provided for at least one (timed) minute twice daily (morning and evening) for 12 weeks.
  Interventions: Drug: Stannous Fluoride Toothpaste (Parodontax Complete Protection Toothpaste)

INTERVENTIONS:
Drug: Stannous Fluoride Toothpaste (Parodontax Complete Protection Toothpaste) — Toothpaste containing 0.454 percent (%) weight by weight (w/w) SnF2.
  Arms: Toothpaste/Mouthwash (SnF2 Toothpaste followed by CPC Mouthwash)
Drug: CPC Mouthwash (Parodontax Active Gum Health Mouthwash) — Mouthwash containing 0.07% w/w CPC.
  Arms: Toothpaste/Mouthwash (SnF2 Toothpaste followed by CPC Mouthwash)
Drug: Regular Fluoride Toothpaste (Crest Cavity Protection) — Toothpaste containing 0.243% w/w sodium fluoride.
  Arms: Negative Control Toothpaste (Sodium Fluoride Toothpaste)
Drug: Stannous Fluoride Toothpaste (Parodontax Complete Protection Toothpaste) — Toothpaste containing 0.454% w/w SnF2.
  Arms: Reference Toothpaste (SnF2 Toothpaste)

SUMMARY:
The aim of this study is to assess the ability of a marketed Cetylpyridinium Chloride (CPC) mouthwash alongside a marketed Stannous Fluoride (SnF2) toothpaste in improving gingival health and reducing plaque accumulation, compared to the use of a regular fluoride toothpaste alone in participants with clinically measurable plaque-induced gingivitis.

DETAILED DESCRIPTION:
This will be a single center, 12-week, randomized, controlled, examiner-blind, 3-treatment arm, parallel group, stratified (by sex [male/female]) study to evaluate the efficacy of using the SnF2 toothpaste/CPC mouthwash twice daily in reducing gingivitis and plaque accumulation in a population with clinically measurable levels of gingivitis. The clinical efficacy of the commercially available SnF2 toothpaste/CPC mouthwash will be compared with that of a commercially available, regular fluoride toothpaste with no known anti-gingivitis nor anti-plaque efficacy properties (negative control). This study will also explore whether a CPC mouthwash used with a SnF2 toothpaste could provide benefits in plaque accumulation reduction and gingival health improvement over the sole use of SnF2 toothpaste (reference product). Sufficient participants will be screened to randomize approximately 198 participants (approximately 66 per group) to ensure approximately 180 evaluable participants (approximately 60 per group) complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant is of either sex and any gender who, at the time of screening, is at least 18 years old, inclusive.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* Participant oral health that meets all the following:

AT SCREENING (Visit 1):

1. Participant with at least 20 natural, permanent teeth.
2. Participant with at least 40 evaluable surfaces for MGI, BI, and TPI.
3. A participant with plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by a gross visual examination at the Screening Visit.

AT BASELINE (Visit 2; Prior to Dental Prophylaxis):

1. A participant with 10% - 30% bleeding sites.
2. A participant with mean interproximal whole mouth TPI score >=1.5.

Exclusion Criteria:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a Haleon employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant who has any other clinical serious or unstable conditions (example, cardiovascular diseases, diabetes, liver disorders, and kidney disorders) which could have affected study outcomes and/or participant safety.
* A participant who is a pregnant female (self-reported) or intending to become pregnant over the duration of the study.
* A female participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* A participant who is a current smoker or an ex-smoker (including vaping) who stopped within 6 months of Screening.
* A participant who is using smokeless forms of tobacco (example, chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant who is diagnosed xerostomia or is taking any medication that in the view of the investigator is causing xerostomia.
* A participant who has a medical condition which could have directly influenced gingival bleeding (example, type 2 diabetes).
* A participant who has a bleeding disorder that could have affected study outcomes and/or participant safety.
* A participant who has a recent history (within the last year) of alcohol or other substance abuse.
* A participant who has a severe oral condition (example, acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/examiner if they participate in the study.
* Presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush.
* Medication exclusions: At screening (Visit 1):

  1. A participant using any antibiotic medication within 4 weeks prior to screening or at any time during the study.
  2. A participant currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition.
  3. A participant currently taking a systemic medication (example, anti-inflammatory, anticoagulant, immunosuppressants) or traditional/ herbal remedy which, in the opinion of the Investigator, could affect plaque/ gingival condition (example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  4. A participant who has used an antibacterial dentifrice or mouthwash (example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, within 4 weeks prior to screening.
* Medication exclusions: At Baseline (Visit 2):

  1. A participant who has taken (in the previous 4 weeks), any antibiotics.
  2. A participant who has taken (in the previous 4 weeks) a systemic medication (example, anti-inflammatory, anti-coagulant, immunosuppressants) or traditional/ herbal remedy (example, ibuprofen, aspirin, warfarin, cyclosporin, phenytoin, calcium channel blockers).
  3. A participant who has used an antibacterial dentifrice or mouthwash (example, chlorhexidine) or any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, in the period between Screening and the Baseline visit.
* Periodontal exclusions:

  1. A participant who has more than three tooth sites with probing pocket depth >= 4 mm.
  2. A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
  3. A participant who has gingivitis, which in the opinion of the investigator, is not expected to respond to treatment with an over the counter (OTC) dentifrice.
* Dental Exclusions:

  1. A participant who has active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  2. A participant who has dentures (partial or full).
  3. A participant who has an orthodontic appliance (bands, appliances, or fixed/removable retainers).
  4. A participant who received orthodontic therapy within 3 months of Screening.
  5. A participant who has numerous restorations in a poor state of repair.
  6. A participant who has any dental condition (example, overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they participate in the study.
  7. A participant who has had dental prophylaxis within 12 weeks of Screening.
  8. A participant who has had teeth bleaching within 12 weeks of Screening.
  9. A participant who has high levels of extrinsic stain or calculus deposits, in the opinion of the investigator, that could have interfered with plaque assessments.
* A participant who has previously been enrolled in this study.
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Overall Number of Bleeding Sites (NBS) at Week 12 (Toothpaste/Mouthwash versus [vs.] Negative Control Toothpaste) | Week 12
  Gingival bleeding will be assessed according to the expanded bleeding index (EBI), by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.

SECONDARY OUTCOMES:
Interproximal NBS at Week 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Overall NBS at Week 6 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Interproximal NBS at Week 6 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Overall Mean Bleeding Index (Bl) at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0=no bleeding after 30 seconds; 1=bleeding observed within 30 seconds of probing; 2=bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Interproximal Mean BI at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0=no bleeding after 30 seconds; 1=bleeding observed within 30 seconds of probing; 2=bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Overall Mean Modified Gingival Index (MGI) at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth (second permanent molar to second permanent molar in each arch) and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation; 1=Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit; 2=Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit; 3=Moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit; 4=Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Interproximal Mean MGI at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth (second permanent molar to second permanent molar in each arch) and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation; 1=Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit; 2=Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit; 3=Moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit; 4=Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Overall Mean Turesky Plaque Index (TPI) at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  The TPI will be used to assess plaque on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores will be recorded buccally/labially (distal, body, mesial sites) and three scores lingually/palatally (distal, body, mesial sites) and mean will be calculated. The plaque will first be disclosed using a plaque disclosing dye solution and the disclosed plaque will be scored on a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin, continuous band of plaque (up to 1 millimeter [mm]) at the cervical margin, 3= Band of plaque wider than 1 mm but covering less than (<)1/3 of the tooth surface, 4= Plaque covering greater than or equal to (>=) 1/3 but < 2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Interproximal Mean TPI at Weeks 6 and 12 (Toothpaste/Mouthwash vs. Negative Control Toothpaste) | Week 6 and Week 12
  The TPI will be used to assess plaque on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores will be recorded buccally/labially (distal, body, mesial sites) and three scores lingually/palatally (distal, body, mesial sites) and mean will be calculated. The plaque will first be disclosed using a plaque disclosing dye solution and the disclosed plaque will be scored on a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin, continuous band of plaque (up to 1 mm) at the cervical margin, 3= Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4= Plaque covering >= 1/3 but < 2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Overall NBS at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Interproximal NBS at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing. The NBS for each participant will be calculated as the number of evaluable tooth sites (having two-thirds of the natural tooth surface gradable for the assessment) with bleeding observed immediately on probing or within 30 seconds of probing.
Overall Mean BI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0=no bleeding after 30 seconds; 1=bleeding observed within 30 seconds of probing; 2=bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Interproximal Mean BI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  Gingival bleeding will be assessed according to the EBI, by inserting a periodontal probe into the gingival crevice and sweeping from distal to mesial around the tooth at an approximate angle of 60 degrees, while in contact with the sulcular epithelium. Each of six gingival areas (distobuccal, midbuccal, mesiobuccal, distolingual, midlingual, and mesiolingual) around each tooth will be assessed. Presence/absence of gingival bleeding will be assessed for 30 seconds after probing and scored on a 3-points scale ranging from 0 to 2, where 0=no bleeding after 30 seconds; 1=bleeding observed within 30 seconds of probing; 2=bleeding observed immediately on probing. Mean BI will be calculated by taking the average over all tooth sites assessed for a participant. Lower score indicates improvement in the symptoms.
Overall Mean MGI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth (second permanent molar to second permanent molar in each arch) and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation; 1=Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit; 2=Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit; 3=Moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit; 4=Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Interproximal Mean MGI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  The MGI assessment is a non-invasive evaluation which focuses on the visual symptoms of gingivitis (for example, redness, texture, edema). MGI will be assessed on the buccal and lingual marginal gingiva and interdental papillae of all scorable teeth (second permanent molar to second permanent molar in each arch) and scored on a 5-point scale ranging from 0 to 4, where 0=Absence of inflammation; 1=Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit; 2=Mild inflammation; criteria as 1 but involving the entire marginal or papillary gingival unit; 3=Moderate inflammation; glazing, redness, edema, and/or hypertrophy of the marginal or papillary gingival unit; 4=Severe inflammation; marked redness, edema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower score indicates improvement in the symptoms.
Overall Mean TPI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  The TPI will be used to assess plaque on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores will be recorded buccally/labially (distal, body, mesial sites) and three scores lingually/palatally (distal, body, mesial sites) and mean will be calculated. The plaque will first be disclosed using a plaque disclosing dye solution and the disclosed plaque will be scored on a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin, continuous band of plaque (up to 1 mm) at the cervical margin, 3= Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4= Plaque covering >= 1/3 but < 2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.
Interproximal Mean TPI at Weeks 6 and 12 (Reference Toothpaste vs. Negative Control Toothpaste) | Week 6 and Week 12
  The TPI will be used to assess plaque on the facial and lingual surfaces of each scorable tooth (second molar to second molar). Three scores will be recorded buccally/labially (distal, body, mesial sites) and three scores lingually/palatally (distal, body, mesial sites) and mean will be calculated. The plaque will first be disclosed using a plaque disclosing dye solution and the disclosed plaque will be scored on a 6-point scale ranging from 0 to 5, where 0=No plaque, 1=Separate flecks of plaque at the cervical margin, 2=Thin, continuous band of plaque (up to 1 mm) at the cervical margin, 3= Band of plaque wider than 1 mm but covering <1/3 of the tooth surface, 4= Plaque covering >= 1/3 but < 2/3 of the tooth surface, 5= Plaque covering >= 2/3 of the tooth surface. Lower score indicates improvement in the symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Salus Research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trialregister@haleon.com.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.